CLINICAL TRIAL: NCT01498640
Title: Retreatment of Recurrent Contractures in Joints Effectively Treated With AA4500 (Collagenase Clostridium Histolyticum [XIAFLEX®/XIAPEX®]) in an Auxilium-sponsored Phase 3 Study in the United States, Australia, and Europe
Brief Title: Retreatment of Recurrent Dupuytren's Contractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-862
Record Dates: First submitted 2011-12-17; First posted 2011-12-23 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Dupuytren's Disease
Keywords: XIAFLEX; XIAPEX; Dupuytren's disease; contracture
MeSH Terms: conditions — Dupuytren Contracture; Contracture | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XIAFLEX/XIAPEX MP Joint (Experimental): Up to 3 injections of collagenase clostridium histolyticum 0.58 mg in the metacarpophalangeal (MP) joint cord
  Interventions: Biological: Collagenase clostridium histolyticum
- XIAFLEX/XIAPEX PIP Joint (Experimental): Up to 3 injections of collagenase clostridium histolyticum 0.58 mg in the proximal interphalangeal (PIP) joint cord
  Interventions: Biological: Collagenase clostridium histolyticum

INTERVENTIONS:
Biological: Collagenase clostridium histolyticum — up to three 0.58 mg injections
  Other Names: XIAFLEX; XIAPEX; AA4500

SUMMARY:
The objectives of this study are to assess the safety and efficacy of AA4500 in the retreatment of recurrent contractures in joints that were effectively treated with AA4500 in a previous Auxilium-sponsored Phase 3 study.

DETAILED DESCRIPTION:
Open-label, Phase 4 study in subjects who are currently participating in the long-term follow-up study (ie, AUX-CC-860) in the United States, Australia, or Europe and who have recurrence of contracture (ie, joint contracture increases by at least 20 degrees compared with the Day 30 value after the last injection in a Phase 3 Auxilium-sponsored study and a palpable cord present) in a joint that was effectively treated (ie, reduction in contracture to 5 degrees or less 30 days after the last injection) with AA4500 in a Phase 3 Auxilium-sponsored study.

Subjects who experience recurrence of contracture in one or more effectively treated joints may be enrolled in this retreatment study after the investigator determines subject eligibility and after informed consent has been obtained. The investigator will treat the cord affecting the recurrent joint with up to three injections. Only one recurrent joint will be treated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Be currently participating in the AUX-CC-860 follow-up study
3. Have at least one joint with all of the following:

   * The joint was effectively treated (had a correction to 5 degrees or less at the Day 30 evaluation after the last injection of AA4500) in a previous Auxilium Phase 3 study
   * The effectively treated joint has an increase in contracture of at least 20 degrees compared with the Day 30 value after the last injection of AA4500 in a previous Auxilium Phase 3 study
   * A palpable cord is present in the joint to be treated
4. Be able to comply with the study visit schedule as specified in the protocol

Exclusion Criteria:

1. Is a pregnant or lactating female or female intending to become pregnant during the study
2. Has hypersensitivity to AA4500 or any of the AA4500 excipients
3. Is currently receiving or plans to receive anticoagulant medication or has received anticoagulant medication (except for equal to or less than 150 mg aspirin daily and over-the-counter nonsteroidal antiinflammatory drugs [NSAIDs]) within 7 days before injection of AA4500

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, MPPH, Study Director — Endo Pharmaceuticals
Locations (13):
- United States (7):
  - HOPE Research Institute, Phoenix, Arizona
  - Rockford Orthopedic Associates, Rockford, Illinois
  - The Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Marquette General Health System, Marquette, Michigan
  - East River Professional Building, New York, New York
  - Health Reserarch Institute, Oklahoma City, Oklahoma
  - Hand Microsurgery and Reconstructive Orthopaedics, Erie, Pennsylvania
- Australia (3):
  - Peninsula Private Hospital, Kippa-Ring, Queensland
  - AusTrials Sherwood, Sherwood, Queensland
  - Emeritus Research, Malvern East, Victoria
- Uppsala Akademiska University Hospital, Uppsala, SE, Sweden
- United Kingdom (2):
  - Pulvertaft Hand Center, Derby, GB
  - Newcastle Upon Tyne Hospitals, Newcastle, GB

RESULTS

PARTICIPANT FLOW:
Groups:
- XIAFLEX/XIAPEX: XIAFLEX/XIAPEX: up to three 0.58 mg injections
Period: Overall Study
Arm/Group | XIAFLEX/XIAPEX
Started | 52
Completed | 47
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
  Australia | 21
  United Kingdom | 4
  Sweden | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Clinical success defined as reduction in fixed-flexion contracture to less than or equal to 5 degrees 30 days after the last injection of AA4500
Time Frame: 30 days after last injection
Population: Efficacy assessment based on modified intent-to-treat (mITT) population which includes all enrolled subjects who received at least 1 AA4500 injection to the treated joint and had at least 1 post-injection efficacy measure
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 31 | 20
percentage of particpants | 64.5 [45.37 to 80.77] | 45.0 [23.06 to 68.47]

2. Primary Outcome: Percent Change From Baseline in Degree of Contracture
Description: Change in fixed-flection contracture measured in degrees where a decrease of 100% would correspond to a reduction in contracture to 0 degrees
Time Frame: Baseline and 30 days after last injection
Population: Efficacy assessment based on mITT population which includes all enrolled subjects who received at least 1 AA4500 injection to the treated joint and had at least 1 post-injection efficacy measure
Measure: Mean (Standard Deviation); unit: percentage of contracture change
Groups:
- XIAFLEX/XIAPEX MP Joint: Up to 3 injections of collagenase clostridium histolyticum 0.58 mg in the MP joint cord
- XIAFLEX/XIAPEX PIP Joint: Up to 3 injections of collagenase clostridium histolyticum 0.58 mg in the PIP joint cord
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 31 | 20
percentage of contracture change | 83.24 (24.275) | 69.10 (26.776)

3. Primary Outcome: Change in Range of Motion
Description: Range of motion defined as difference between full flexion angle and full extension angle expressed in degrees
Time Frame: Baseline and 30 days after last injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 31 | 20
degrees | 31.4 (17.52) | 26.8 (17.39)

4. Secondary Outcome: Physician Global Assessment of Improvement
Description: Physician global assessment of change (improvement) in subject's Dupuytren's contracture
Time Frame: 30 days after last injection
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 31 | 20
participants
  Very much improved | 18 | 12
  Much improved | 11 | 5
  Minimally improved | 0 | 2
  No change | 1 | 1
  Minimally worse | 0 | 0
  Much worse | 0 | 0
  Very much worse | 0 | 0
  Not done | 1 | 0

5. Secondary Outcome: Subject Global Assessment of Satisfaction
Description: Subject global assessment of overall treatment satisfaction
Time Frame: 30 days after last injection
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 31 | 20
participants
  Very satisfied | 20 | 10
  Quite satisfied | 9 | 5
  Neither satisfied nor dissatisfied | 1 | 2
  Quite dissatisfied | 0 | 1
  Very dissatisfied | 0 | 0
  Not done | 1 | 2

6. Secondary Outcome: Recurrence of Contracture
Description: Recurrence of contracture in the joint at day 365 that was successfully treated 30 days after last injection assessed. Recurrence was defined as 20 degree or greater increase of contracture of the treated joint at day 365 or medication intervention of the treated joint between the 2 time points.
Time Frame: Day 365
Population: Efficacy assessment based on mITT population which includes all enrolled subjects who received at least 1 AA4500 injection to the treated joint and had at least 1 post-injection efficacy measure; only joints that were successfully treated (reduction in contracture to 5 degrees or less) 30 days after last injection were assessed
Measure: Number; unit: joints
Units Other Than Participants: Joints
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 29
Number analyzed (Joints) | 29
joints | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | XIAFLEX/XIAPEX
Serious Adverse Events (participants affected / at risk) | 4/52
Other Adverse Events (participants affected / at risk) | 44/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIAFLEX/XIAPEX (N=52)
Cerebellar infarction (Nervous system disorders) | 1 (1) — Resulted in death
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIAFLEX/XIAPEX (N=52)
Oedema peripheral (General disorders) | 32 (41)
Contusion (Injury, poisoning and procedural complications) | 23 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (22)
Injection site pain (General disorders) | 10 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (13)
Injection site haematoma (General disorders) | 8 (12)
Lymphadenopathy (Blood and lymphatic system disorders) | 8 (8)
Skin laceration (Injury, poisoning and procedural complications) | 7 (7)
Injection site pruritus (General disorders) | 5 (5)
Injection site swelling (General disorders) | 5 (9)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other